CLINICAL TRIAL: NCT04506697
Title: Study of Remote Monitoring of Urination Dynamics
Brief Title: Remote Monitoring of Uroflowmetry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Institute for Digital Medicine (WisDM) (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CM-001
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with LUTS (Experimental): Patients who are indicated for uroflowmetry
  Interventions: Procedure: Uroflowmetry

INTERVENTIONS:
Procedure: Uroflowmetry — The patient is given a portable uroflowmeter for performing uroflowmetry at home, and the NetHealth app is installed on his smartphone. The patient registers his account in the app. A personal uroflowmeter is paired with the patient's smartphone using the installed app via a Bluetooth connection. The investigator trains the patient how to use the app and how to conduct uroflowmetry at home. The patient within 1 day (24 hours) at home performs uroflowmetry during all urination, including night urination.

SUMMARY:
The aim of the study is to assess the possibility of using remote monitoring of urination.

ELIGIBILITY:
Inclusion Criteria:

1. Men over 18 years old.
2. The patient has performed uroflowmetry according to indications in the hospital no later than 7 days before the planned inclusion in the trial.
3. Qmax = or <15 ml / sec.
4. The patient has a smartphone (with Android 4.0 and higher, iOS 10.0 and higher) with Internet access

Exclusion Criteria:

1. A patient with emergency conditions requiring surgical treatment
2. Intellectual and cognitive abilities of the patient that do not allow him to follow the doctor's instructions and make it difficult to use the smartphone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Uroflowmetry during 24 hours | 1 day
  Registration of remote uroflowmetry using portable uroflowmeter during 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No